CLINICAL TRIAL: NCT00970788
Title: A Pilot Study of Using Video Images in Advance Care Planning in Malignant Glioma Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Foundation for Informed Medical Decision Making (Other)
Responsible Party: Principal Investigator, Angelo E. Volandes, MD, Faculty, Massachusetts General Hospital
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2008-P-000826/6
Record Dates: First submitted 2009-08-07; First posted 2009-09-02 (Estimated); Last update posted 2012-05-01 (Estimated); Status verified 2012-04

CONDITIONS: Advanced Brain Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- verbal group (No Intervention): Verbal description of goals of care.
- Video group (Experimental): Video decision aid.
  Interventions: Behavioral: Video intervention

INTERVENTIONS:
Behavioral: Video intervention — Video of goals of care
  Arms: Video group

SUMMARY:
A randomized controlled trial of a video decision aid in 50 patients with advanced brain cancer.

DETAILED DESCRIPTION:
A randomized controlled trial of a video decision aid in 50 patients with advanced brain cancer. Subjects will have three options for their goals of care: life prolonging care, basic medical care, or comfort care.

ELIGIBILITY:
Inclusion Criteria:

* Advanced brain cancer
* English Speaking
* Able to provide informed consent

Exclusion Criteria:

* Folstein mini mental status score of 23 or less

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2008-07; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

PRIMARY OUTCOMES:
end of life preference at time of interview | 5 minutes after survey

SECONDARY OUTCOMES:
uncertainty regarding end of life preference at time of interview | 5 minutes after survey
knowledge of end of life preference at time of interview | 5 minutes after survey

CONTACTS AND LOCATIONS:
Overall Officials: Angelo Volandes, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- MGH, Boston, Massachusetts, United States